CLINICAL TRIAL: NCT05826756
Title: Project PEER: Understanding the Lung Cancer Patient ExperiEnce in the Real-World Setting
Acronym: PEER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LUNGevity Foundation (Other)
Collaborators: Amgen (Industry); AstraZeneca (Industry); Blueprint Medicines Corporation (Industry); Boehringer Ingelheim (Industry); Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry); G1 Therapeutics, Inc. (Industry); Genentech, Inc. (Industry); Janssen, LP (Industry); Jazz Pharmaceuticals (Industry); Merck Sharp & Dohme LLC (Industry); Novartis (Industry); Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: LUNGevity-2020-01
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer Patients; Caregivers
Keywords: Lung cancer; Patient; Caregiver; Smoker; Non-smoker; Tobacco use; Tobacco exposure; Biomarker; Non-small cell lung cancer (NSCLC); Small cell lung cancer (SCLC); Quality of life; Treatment
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Individuals who have been diagnosed with lung cancer. Individuals with all stages of lung cancer and individuals who have reached no evidence of disease (NED).
  Interventions: Other: There are no interventions in this study. All participants complete online surveys.
- Caregivers: Family and friends who provide care for someone who has been diagnosed with lung cancer
  Interventions: Other: There are no interventions in this study. All participants complete online surveys.

INTERVENTIONS:
Other: There are no interventions in this study. All participants complete online surveys. — There are no interventions in this study. All participants complete online surveys.
  Other Names: Other

SUMMARY:
LUNGevity Foundation, a non-profit lung cancer organization, wants to learn about living with lung cancer from the point of view of people with lung cancer and their family and friends who provide care. To do this, we have an online study designed to better understand how treatments people living with lung cancer receive impact their quality of life. Participants will complete surveys once a month for 12 months.

What does participation involve?

1. Emailing the study team to learn more and get access to the study website.
2. Once a month for 12 months you will receive a survey by email.
3. Complete these surveys on a smartphone, tablet, or computer at your convenience and receive an e-gift card for your time.

DETAILED DESCRIPTION:
PEER is an international study, that is Institutional Review Board (IRB) approved and General Data Protection Regulation (GDPR) compliant.

The study objective is to collect longitudinal data to facilitate a rigorous understanding of the diagnostic and treatment experiences of people diagnosed with lung cancer and to identify determinants of treatment heterogeneity. Study data will be used to understand the diagnostic and treatment pathways, explore patient-experience data in different domains (financial impact/quality of life/symptoms) and test the hypothesis that different classes of therapies (chemotherapy/ immunotherapy/ targeted therapy/ surgery/ radiation) impact patient experience (eg., physical function).

Study participants will consent and register for the study and complete an initial baseline survey. They will then be followed for 12 months and receive a monthly survey (11 surveys in total) via email. The development of the surveys was guided by input from patients, clinicians, FDA experts, and incorporates questions from existing patient-reported outcomes (PRO) measures.

Summarized study results will also be posted on LUNGevity's website. External researchers will be able to apply to have limited access to de-identified data.

ELIGIBILITY:
Inclusion Criteria:

* Adults with self-reported lung cancer diagnosis or caregiver of someone with a self-reported lung cancer diagnosis (patient has to be alive)
* Ability to read and answer questions in English
* Access and ability to use a computer or other internet-connected device

Exclusion Criteria:

* Younger than 18
* Healthcare providers and healthcare professionals who provide care to lung cancer patients except for those who are themselves a patient or a caregiver to a loved one.
* Not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have been diagnosed with lung cancer and family and friends who care for someone with a lung cancer diagnosis. PEER is an international study, so participants can live anywhere as long as they meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Explore guideline concordant care | From baseline and assessed monthly up to end of study (up to approximately 12months)
  Patient-reported treatments will be explored in relation to other clinical data provided (e.g., biomarker presence) and the National Comprehensive Cancer Network (NCCN) guidelines for those clinical characteristics at the time of treatment.
Explore patient-reported functioning, symptoms, side effects and overall quality of life | From baseline and assessed monthly up to end of study (up to approximately 12months)
  Patterns based on disease staging and treatment class will be explored using the European Organisation for Research and Treatment of Cancer Quality of Life 30-item questionnaire (EORTC QLQ-C30), the Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ), and a side effect questionnaire to explore these patient-reported outcomes.
  Scores for the EORTC QLQ-C30 are transformed so that for each subscale the range is 0-100. For functioning subscales, higher scores indicate better functioning, and for symptoms higher scores indicate more symptom burden. Scores for the NSCLC-SAQ range from 0-20, with higher scores indicating more severe symptomology.
Explore impacts of different classes of therapies | From baseline and assessed monthly up to end of study (up to approximately 12months)
  Test whether different classes of therapies (e.g., chemotherapy/ immunotherapy/ targeted therapy/ surgery/ radiation) impact patient experience (e.g., side effects, functioning). Both within and between patient experiences will be investigated. Results from Project PEER will be compared currently existing clinical trial data.

OTHER OUTCOMES:
Impact of the pandemic on access to treatment | Baseline survey - Temporary COVID-19 module
  Exploratory descriptive analyses to understand the concerns participants who enrolled in 2020 and 2021 experienced with respect to their treatment and COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Upal Basu Roy, PhD, MPH, Principal Investigator — LUNGevity Foundation
Locations (1):
- LUNGevity Foundation, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT05826756/Prot_SAP_000.pdf